CLINICAL TRIAL: NCT05668312
Title: Effects of Tele-prehabilitation on Clinical and Muscular Recover in Patients Waiting for Knee Replacement: a Randomized Controlled Trial
Brief Title: Effects of Tele-prehabilitation in Patients Waiting for Knee Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tele-prehabilitation
Record Dates: First submitted 2022-11-22; First posted 2022-12-29 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Tele-prehabilitation; Prehabilitation; Virtual Reality; Advanced technologies; Knee osteoarthritis; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: The forty-eight subjects undergoing prehabilitation will be randomly allocated to one of the two possible intervention arms (tele-prehabilitation or standard prehabilitation). The twenty healthy young subject will not undergo any prehabilitation and will not be allocated to one of the two prehabilitation arms.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TELE-pre group (Experimental): Subjects in the TELE-prehabilitation group receive remote prehabilitation using advanced technologies.
  Interventions: Other: Tele-prehabilitation
- Control group (Active Comparator): The control group is composed by the Con-O (Control Older) group and the Con-Y (Control Young) group. In the Con-O group (n=24) subjects receive home-based prehabilitation using a printed booklet; in the Con-Y group (n=20) subjects do not receive any prehabilitation program.
  Subjects in the Con-Y group will be recruited from patients waiting for anterior cruciate ligament reconstruction, thus they will be only assessed with muscular biopsy and blood sampling.
  Interventions: Other: Standard prehabilitation

INTERVENTIONS:
Other: Tele-prehabilitation — Preoperative tele-rehabilitation using a virtual reality system.
  Arms: TELE-pre group
Other: Standard prehabilitation — Preoperative home-based rehabilitation delivered with a printed booklet for the Con-O subjects and no intervention for the Con-Y subjects.
  Arms: Control group

SUMMARY:
After knee arthroplasty rehabilitation is fundamental to patient's functional recovery, but in recent years there has been a growing interest in the possibility to prepare patients for surgery through a "prehabilitation" program. This two-parallel groups randomized clinical trial aims at evaluating the effects of a preoperative rehabilitation programme carried out at patient's home using advanced technologies, on subjects waiting for knee replacement. In particular, the primary objective of this study is to assess the superiority of a tele-prehabilitation programme compared to standard prehabilitation (remotely delivered with a booklet) in determining an improvement in lower limb function, as measured by the Western Ontario and McMaster Universities Osteoarthritis Index questionnaire, at the end of the programme. This study also aims at assessing possible differences between groups in muscle function, pain, autonomy in the activity of daily living, adherence to treatment and patients' satisfaction with the prehabilitation modality. Through the analysis of quadriceps muscle and blood samples, we will also evaluate possible changes in the expression of specific markers that the prehabilitation programme may be able to determine at muscle level. Both the intervention and the control groups will perform a prehabilitation program in the 6 weeks just before surgery. The program will include therapeutic exercises and educational contents. Subjects in the tele-prehabilitation group will receive a tablet with two accelerometers and a balance board for the remote execution of the program, while the control group will receive the same intervention through a booklet. Subjects recruited will be assessed at 5 timepoints: before starting the prehabilitation program, the day of surgery, 7± 2 and 15 ± 2 days after surgery, 3 months ± 7 days after surgery.

DETAILED DESCRIPTION:
Based on the existing literature, we expected to observe an effect size of 0.8 in WOMAC (primary outcome) between groups at the end of the tele-prehabilitation program. Therefore, considering a test power of 80% and an alpha error of 5%, we have computed a sample size of 48 subjects, 24 for each group (taking into account a possible drop-out rate of 15-20%).

Twenty healthy young subjects (10 males and 10 females) will be also recruited only for muscle and blood samples collection, that will be used as benchmarks for the intervention and control groups analyses (they will no undergo any prehabilitation program).

The recruited subjects will be randomly allocated (with a 1:1 ratio randomization list) in the tele-prehabilitation or in the control groups. During the 6 weeks just before surgery, both groups will perform 5 sessions a week of the same home-based prehabilitation program. Each session is planned as follow: 5 minutes of warm-up, 30 minutes of work (mobility, strengthening and balance exercises) and 5 minutes of cool-down.

In details, for each session subjects will perform the following exercises:

1. Warm-up (about 5 minutes)

   1. Knee bending and extension in lying position;
   2. Knee extensions while sitting;
   3. Get on tiptoes in standing position;
   4. March on site.
2. Working phase (about 30 minutes)

   1. Hip bending keeping the knee extended in lying position;
   2. Hip motion in space planes (imagining of drawing numbers with the tiptoe);
   3. Hip abduction keeping the knee extended side lying;
   4. Knee bending and hip extension in standing position;
   5. Half squat;
   6. Half lateral lunge;
   7. Monopodalic standing;
   8. Tandem walking;
   9. Weight shifting on unstable surface.
3. Cool-down (about 5 minutes)

   1. Free walk;
   2. Leg swings while sitting.

Subjects of both groups will also have to read, once a week, an educational content (digital for the tele-prehabilitation group, printed for the control one) dealing with:

* Information about knee osteoarthritis and replacement;
* Post-operative symptoms, what to expect;
* Advices for home organization after surgery;
* Healthy life style: physical activity, nutrition and sleep;
* Advices for maintaining progresses;
* Motivational intervention.

The tele-prehabilitation program will be delivered using the following devices (Khymeia, Padova, Italy -Khymeia - e-health innovation):

* TeleCockpit, a workstation used by the clinician to manage remotely patient's home device, interact real-time or check the adherence to treatment;
* VRRS Home Tablet, with an uploaded mobile application for the exercises execution at home;
* VRRS Khymu, two accelerometers for patient's interaction with the virtual reality system during knee motion;
* VRRS Balance, a balance board for patient's interaction with the virtual reality system during centre-of-mass motion.

The exercise volume of the "work" section of the prehabilitative session will increase during the 6 weeks according to patient's symptoms. This progression will be based on the score, measured at the end of each workout, obtained at the Borg CR-10 scale self-administered by the patient at the end of each session. A score below 5 indicates the need to increase the workload in the next session. The progression of the working volume will be considered and eventually managed weekly by the clinician in charge, for the intervention group connecting to the patient's device with the TeleCockpit workstation, and for the control group by communicating the changes in the prescription details with a phone call.

ELIGIBILITY:
Inclusion Criteria for TELE-pre and Con-O groups (also previous information are valid only for these groups):

* Scheduled unilateral total knee replacement surgery according to Fast-Track pathway;
* Preoperative criteria for home discharge;
* At least one person cohabitant;
* Familiarity with tablet/computer use and Internet access;
* Informed consent signature.

Inclusion Criteria for Con-Y group:

* Both sexes of any ethnicity;
* Age between 18 and 35 years;
* Scheduled Anterior Cruciate Ligament reconstruction surgery;
* Body Mass Index ≤ 30.

Exclusion Criteria for TELE-pre and Con-O groups:

* Scheduled surgery for knee revision arthroplasty;
* Lower limbs surgery in the previous 6 months;
* Lower limbs fractures in the previous 6 months;
* Congenital or post-traumatic knee morphologic alterations;
* Rehabilitation treatments in the previous 6 months focused on the interested knee functional recovery;
* Ongoing neurological or oncological diseases;
* HIV, HCV, HBV, TPHA infection;
* Cognitive impairment;
* Known local anaesthetics allergic reactions;
* Ongoing non-suspendable anticoagulant therapies;
* Known muscular diseases.

Exclusion Criteria for Con-Y group:

* Body Mass Index > 30;
* Ongoing oncological diseases;
* Sampling area infection;
* HIV, HCV, HBV, TPHA infection;
* Known neuromuscular/muscular diseases;
* Ongoing non-suspendable anticoagulant therapies,
* Female subjects in pregnancy status or breastfeeding.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at 6/7 weeks | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1).
  The WOMAC questionnaire is a self-administrated health status measure for pain, stiffness and function assessment in patients with hip or knee osteoarthritis. It is composed by 24 items and uses a 5-point Likert scale (from 0 to 4).

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  The WOMAC questionnaire is a self-administrated health status measure for pain, stiffness and function assessment in patients with hip or knee osteoarthritis. It is composed by 24 items and uses a 5-point Likert scale (from 0 to 4).
Oxford Knee Score (OKS) | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  The OKS is a self-administrated questionnaire assessing symptoms and function in patients undergoing knee replacement. It is composed by 12 items and uses a 5-point Likert scale.
Numeric Pain Rating Scale (NPRS) | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  The NPRS is an 11-point scale from 0 to 10 assessing pain. "0" is "no pain", "10" is "the most intense pain imaginable".
Short Form-12 | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  The Short Form-12 is questionnaire for health assessment, composed by 12 items, which can be self-administrated or completed through an interview. An algorithm is used to obtain the final composite score.
International Physical Activity Questionnaire (IPAQ) | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  The IPAQ is a 9-item self-reported measure of physical activity. Adding up the week minutes of walking, moderate-intensity activity and vigorous-intense activity, multiplied per specific coefficients, the questionnaire estimate the overall Metabolic Equivalent of Task.
Sit-to-stand test | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  The subject is asked to stand-up and sit-down on a chair, standardized in size, for 5 consecutive times as much faster as he can. Time (in seconds) to complete the task is representative of the lower limb strength.
Knee extensor and flexors maximal strength assessment | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  Maximal strength will be assessed using a dynamometer and expressed in kilograms (Kg).
Timed Up-and-Go test | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  The subject is asked, starting from seated on a chair, to stand-up, walk 3m, go back to the chair and sit-down. Time (in seconds) to complete the task is representative of the subject's risk of fall.
Knee Range Of Motion | The day of the recruitment (T0); 6/7 weeks after T0, the day of surgery (T1); 7 +/- 2 days after surgery (T2); 15 +/- 2 days after surgery (T3); 90 +/- 7 days after surgery (T4)
  Knee motion in flexion and extension is measured using a goniometer and expressed in degree.
Satisfaction interview | 6/7 weeks after T0.
  This interview is a 6-item self-reported measure of participant's satisfaction about the prehabilitation delivery modality, which uses a 11-point Likert scale.
  This interview has been created ad hoc for this study.
Prehabilitation diary | 6/7 weeks after T0.
  This diary has been created ad hoc to assess participant's adherence to treatment. The measure of adherence is expressed by the total number of sessions reported in the diary.
  It will be used only to assess adherence of the Con-O group.
Muscle metabolism markers | The day of the recruitment (T0); the day of surgery (T1); 90 +/- 7 days after surgery (T4)
  Muscle will be sampled by needle aspiration (for participants belonging to Tele-pre or Con-O groups) or discarded muscle material collection during surgical procedures.
  In collected muscle samples, myosin heavy chain (MHC) isoform distribution will be assessed by SDS-PAGE electrophoresis, while levels of markers as PGC1alpha will be investigated by ELISA or Western Blot. Proteomics analysis will be conducted by LC-MS, using TMT quantification, whereas lipidomics and sphingolipidomics analyses will be conducted by untargeted and targeted LC-MS.
Blood biomarkers | The day of the recruitment (T0); the day of surgery (T1); 90 +/- 7 days after surgery (T4)
  Blood sample will taken according to standard procedures. Levels of proteins or lipids suggested to be potential biomarkers will be investigated in collected sera, by ELISA or MRM-MS.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mangiavini, Principal Investigator — IRCCS Galeazzi - Sant'Ambrogio Hospital; Giuseppe Peretti, Principal Investigator — IRCCS Istituto Clinico San Siro
Locations (2):
- Italy (2):
  - IRCCS Istituto Clinico San Siro, Milan
  - IRCCS Ospedale Galeazzi - Sant'Ambrogio (Coordinator), Milan

REFERENCES:
- [Background] Romanini E, Decarolis F, Luzi I, Zanoli G, Venosa M, Laricchiuta P, Carrani E, Torre M. Total knee arthroplasty in Italy: reflections from the last fifteen years and projections for the next thirty. Int Orthop. 2019 Jan;43(1):133-138. doi: 10.1007/s00264-018-4165-7. Epub 2018 Oct 6. PMID 30293141
- [Background] Erivan R, Tardieu A, Villatte G, Ollivier M, Jacquet C, Descamps S, Boisgard S. Knee surgery trends and projections in France from 2008 to 2070. Orthop Traumatol Surg Res. 2020 Sep;106(5):893-902. doi: 10.1016/j.otsr.2020.02.018. Epub 2020 Jun 4. PMID 32507586
- [Background] Hitzl W, Heisinger S, Hobusch GM, Frank K, Cotofana S. Projected numbers of primary total knee replacement in Austria from 2015-2075. Orthopade. 2019 Feb;48(2):144-149. doi: 10.1007/s00132-018-3605-9. PMID 30051278
- [Background] Singh JA, Yu S, Chen L, Cleveland JD. Rates of Total Joint Replacement in the United States: Future Projections to 2020-2040 Using the National Inpatient Sample. J Rheumatol. 2019 Sep;46(9):1134-1140. doi: 10.3899/jrheum.170990. Epub 2019 Apr 15. PMID 30988126
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] L Snell D, Hipango J, Sinnott KA, Dunn JA, Rothwell A, Hsieh CJ, DeJong G, Hooper G. Rehabilitation after total joint replacement: a scoping study. Disabil Rehabil. 2018 Jul;40(14):1718-1731. doi: 10.1080/09638288.2017.1300947. Epub 2017 Mar 23. PMID 28330380
- [Background] Vasta S, Papalia R, Torre G, Vorini F, Papalia G, Zampogna B, Fossati C, Bravi M, Campi S, Denaro V. The Influence of Preoperative Physical Activity on Postoperative Outcomes of Knee and Hip Arthroplasty Surgery in the Elderly: A Systematic Review. J Clin Med. 2020 Mar 31;9(4):969. doi: 10.3390/jcm9040969. PMID 32244426
- [Background] Jette DU, Hunter SJ, Burkett L, Langham B, Logerstedt DS, Piuzzi NS, Poirier NM, Radach LJL, Ritter JE, Scalzitti DA, Stevens-Lapsley JE, Tompkins J, Zeni J Jr; American Physical Therapy Association. Physical Therapist Management of Total Knee Arthroplasty. Phys Ther. 2020 Aug 31;100(9):1603-1631. doi: 10.1093/ptj/pzaa099. PMID 32542403
- [Background] Moyer R, Ikert K, Long K, Marsh J. The Value of Preoperative Exercise and Education for Patients Undergoing Total Hip and Knee Arthroplasty: A Systematic Review and Meta-Analysis. JBJS Rev. 2017 Dec;5(12):e2. doi: 10.2106/JBJS.RVW.17.00015. PMID 29232265
- [Background] Doiron-Cadrin P, Kairy D, Vendittoli PA, Lowry V, Poitras S, Desmeules F. Feasibility and preliminary effects of a tele-prehabilitation program and an in-person prehablitation program compared to usual care for total hip or knee arthroplasty candidates: a pilot randomized controlled trial. Disabil Rehabil. 2020 Apr;42(7):989-998. doi: 10.1080/09638288.2018.1515992. Epub 2019 Jan 13. PMID 30638076
- [Background] Sharif F, Rahman A, Tonner E, Ahmed H, Haq I, Abbass R, Asinger S, Sbai M. Can technology optimise the pre-operative pathway for elective hip and knee replacement surgery: a qualitative study. Perioper Med (Lond). 2020 Nov 16;9(1):33. doi: 10.1186/s13741-020-00166-0. PMID 33292556
- [Background] McDonnell JM, Ahern DP, Ross TD, Gibbons D, Synnott KA, Butler JS. The efficacy of remote virtual care in comparison to traditional clinical visits for elective orthopaedic patients: A meta-analysis of prospective randomised controlled trials. Surgeon. 2022 Jun;20(3):177-186. doi: 10.1016/j.surge.2021.02.008. Epub 2021 Mar 21. PMID 33762159
- [Background] Wang Q, Lee RLT, Hunter S, Chan SW. The effectiveness of internet-based telerehabilitation among patients after total joint arthroplasty: An integrative review. Int J Nurs Stud. 2021 Mar;115:103845. doi: 10.1016/j.ijnurstu.2020.103845. Epub 2020 Dec 6. PMID 33360248
- [Background] Harmelink KEM, Zeegers AVCM, Tonis TM, Hullegie W, Nijhuis-van der Sanden MWG, Staal JB. The effectiveness of the use of a digital activity coaching system in addition to a two-week home-based exercise program in patients after total knee arthroplasty: study protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2017 Jul 5;18(1):290. doi: 10.1186/s12891-017-1647-5. PMID 28679400
- [Background] Correia FD, Nogueira A, Magalhaes I, Guimaraes J, Moreira M, Barradas I, Molinos M, Teixeira L, Tulha J, Seabra R, Lains J, Bento V. Medium-Term Outcomes of Digital Versus Conventional Home-Based Rehabilitation After Total Knee Arthroplasty: Prospective, Parallel-Group Feasibility Study. JMIR Rehabil Assist Technol. 2019 Feb 28;6(1):e13111. doi: 10.2196/13111. PMID 30816849
- [Background] Bell KM, Onyeukwu C, McClincy MP, Allen M, Bechard L, Mukherjee A, Hartman RA, Smith C, Lynch AD, Irrgang JJ. Verification of a Portable Motion Tracking System for Remote Management of Physical Rehabilitation of the Knee. Sensors (Basel). 2019 Feb 28;19(5):1021. doi: 10.3390/s19051021. PMID 30823373
- [Background] Jansson MM, Rantala A, Miettunen J, Puhto AP, Pikkarainen M. The effects and safety of telerehabilitation in patients with lower-limb joint replacement: A systematic review and narrative synthesis. J Telemed Telecare. 2022 Feb;28(2):96-114. doi: 10.1177/1357633X20917868. Epub 2020 Apr 21. PMID 32316837
- [Background] An J, Ryu HK, Lyu SJ, Yi HJ, Lee BH. Effects of Preoperative Telerehabilitation on Muscle Strength, Range of Motion, and Functional Outcomes in Candidates for Total Knee Arthroplasty: A Single-Blind Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Jun 4;18(11):6071. doi: 10.3390/ijerph18116071. PMID 34199913
- [Background] Chughtai M, Shah NV, Sultan AA, Solow M, Tiberi JV, Mehran N, North T, Moskal JT, Newman JM, Samuel LT, Bhave A, Mont MA. The role of prehabilitation with a telerehabilitation system prior to total knee arthroplasty. Ann Transl Med. 2019 Feb;7(4):68. doi: 10.21037/atm.2018.11.27. PMID 30963063
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188
- [Background] Botolfsen P, Helbostad JL, Moe-Nilssen R, Wall JC. Reliability and concurrent validity of the Expanded Timed Up-and-Go test in older people with impaired mobility. Physiother Res Int. 2008 Jun;13(2):94-106. doi: 10.1002/pri.394. PMID 18288773
- [Background] Salaffi F, Leardini G, Canesi B, Mannoni A, Fioravanti A, Caporali R, Lapadula G, Punzi L; GOnorthrosis and Quality Of Life Assessment (GOQOLA). Reliability and validity of the Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index in Italian patients with osteoarthritis of the knee. Osteoarthritis Cartilage. 2003 Aug;11(8):551-60. doi: 10.1016/s1063-4584(03)00089-x. PMID 12880577
- [Background] Padua R, Zanoli G, Ceccarelli E, Romanini E, Bondi R, Campi A. The Italian version of the Oxford 12-item Knee Questionnaire-cross-cultural adaptation and validation. Int Orthop. 2003;27(4):214-6. doi: 10.1007/s00264-003-0453-x. Epub 2003 Apr 2. PMID 12679892
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Kodraliu G, Mosconi P, Groth N, Carmosino G, Perilli A, Gianicolo EA, Rossi C, Apolone G. Subjective health status assessment: evaluation of the Italian version of the SF-12 Health Survey. Results from the MiOS Project. J Epidemiol Biostat. 2001;6(3):305-16. doi: 10.1080/135952201317080715. PMID 11437095
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588
- [Derived] Guida S, Vitale J, Gianola S, Castellini G, Swinnen E, Beckwee D, Gelfi C, Torretta E, Mangiavini L. Effects of tele-prehabilitation on clinical and muscular recovery in patients awaiting knee replacement: protocol of a randomised controlled trial. BMJ Open. 2023 Oct 4;13(10):e073163. doi: 10.1136/bmjopen-2023-073163. PMID 37793919